CLINICAL TRIAL: NCT00285584
Title: Drug Abuse, Depression and Responses to HIV Counseling
Brief Title: Bupropion For Reducing High-Risk Behaviors in Depressed Men Who Have Sex With Men (MSM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIDA-15303-1; R01DA015303 (NIH); DPMC
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: HIV Infections; Depression
Keywords: HIV infection; Depression; Men who have sex with men; Drug abuse
MeSH Terms: conditions — HIV Infections; Depression; Homosexuality; Substance-Related Disorders | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupropion (Active Comparator): Participants in this arm received bupropion.
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Participants in this arm received placebo that looked identical to the active comparator medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion — Participants initially received bupropion, 150 mg, once daily, to be taken in the morning. Dosage was increased to 150 mg twice daily within one month. Return visits were conducted monthly from study Months 1 through 6 to review medication dosage, ascertain side effects and evaluate depression severity. At the end of Moth 6, subjects were tapered to 150 mg/day over a period of 4 - 7 days. The final 150 mg/day dosage of bupropion allowed referral for pharmacotherapy without unblinding subjects or staff regarding bupropion/placebo assignment. Subjects were followed through Month 9 to permit evaluation of the durability of intervention effects.
  Other Names: Brand name of bupropion used in the trial: Wellbutrin SR
  Arms: Bupropion
Drug: Placebo — Participants initially received placebo, 150 mg, once daily, to be taken in the morning. Dosage was increased to 150 mg twice daily within one month. Return visits were conducted monthly from study Months 1 through 6 to review medication dosage, ascertain side effects and evaluate depression severity. At the end of Moth 6, subjects were tapered to 150 mg/day over a period of 4 - 7 days. The final 150 mg/day dosage allowed referral for pharmacotherapy without unblinding subjects or staff regarding bupropion/placebo assignment. Subjects were followed through Month 9 to permit evaluation of the durability of intervention effects.
  Arms: Placebo

SUMMARY:
The primary purpose of this study was to test the whether high-risk, HIV-seronegative persons with mild-to-moderate depression would be more likely to adopt protective behavior change when provided with pharmacotherapy for their depression than when treated with placebo. High-risk behaviors include using illegal drugs and participating in unprotected sexual intercourse. The specific pharmacotherapy used in this study was the anti-depressant, bupropion. The subject population consisted of HIV negative men who have sex with men (MSM) with mild-to-moderate depression.

DETAILED DESCRIPTION:
Depression in men is often masked by high-risk behaviors such as alcohol and drug abuse. Common symptoms among depressed men include feelings of hopelessness and helplessness, irritability, and anger. MSM are among those at highest for HIV acquisition due to high-risk behaviors, including unprotected sexual intercourse and drug abuse. Bupropion is an antidepressant medication commonly used to treat depression. The purpose of this study thus was whether bupropion could help MSM with mild-to-moderate depression reduce their high-risk behaviors.

Participants in this trial were randomly assigned to receive either bupropion or placebo for 6 months. Study visits lasting approximately 2 hours each occurred at Day 0, and at Months 4, 6, and 9; included in these visits were physical examination, testing for HIV and sexually transmitted disease (STD), depression screening, and an interview-administered questionnaire inquiring into sexual activity and drug use. Shorter study visits, lasting 15 - 30 minutes each occurred at Day 15, and Months 1, 2, 4, 5, and 7, and included depression screening and physical exam.

ELIGIBILITY:
Inclusion Criteria:

* Available for at least 9 months, or the duration of the study
* Willing to complete HIV testing and counseling
* History of HIV testing and counseling
* At high risk of HIV infection, indicated by more than one male sexual partner in the 3 months prior to study entry
* Meets criteria for either (a) major depression or dysthymia within a mild-to-moderate level according to standard criteria DSM-IV, or (b) minor depression as defined by one or more of the following symptoms at any time and for any duration during the past 12 months: significant weight loss or gain, or significant decrease or increase in appetite; poor sleep pattern; noticeable irritability or slowness; fatigue or lack of energy; inappropriate feelings of worthlessness or guilt; inability to concentrate; indecisiveness; and recurrent thoughts of death or suicide.

Exclusion Criteria:

* HIV infected
* Sexual intercourse in the 3 months prior to study entry with only one partner, and in a monogamous relationship
* Currently enrolled in another study involving repeated HIV testing and counseling
* Receiving treatment for depression with antidepressant medication for any length of time within the year prior to study entry
* Currently in psychotherapy, psychoanalysis, or any other form of talk therapy for any reason
* Severe depression or at suicidal risk
* No evidence or prior history of depression
* Homicidal or other similar problem that, in the opinion of the investigator, may endanger study staff and participants
* Currently taking monoamine oxidase inhibitors (MAOIs). Participants may be allowed to enroll 14 days after discontinuing use of a MAOI.
* History of seizures
* History or current symptoms of bipolar disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-09; Primary Completion 2004-03 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marmor, PhD, Principal Investigator — Department of Environmental Medicine, New York University
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - New York University School of Medicine, New York, New York

REFERENCES:
- [Background] Thomas SM, Tse DB, Ketner DS, Rochford G, Meyer DA, Zade DD, Halkitis PN, Nadas A, Borkowsky W, Marmor M. CCR5 expression and duration of high risk sexual activity among HIV-seronegative men who have sex with men. AIDS. 2006 Sep 11;20(14):1879-83. doi: 10.1097/01.aids.0000244207.49123.ff. PMID 16954729
- [Background] Marmor M, Hertzmark K, Thomas SM, Halkitis PN, Vogler M. Resistance to HIV infection. J Urban Health. 2006 Jan;83(1):5-17. doi: 10.1007/s11524-005-9003-8. PMID 16736351
- [Background] Halkitis PN, Zade DD, Shrem M, Marmor M. Beliefs about HIV non-infection and risky sexual behavior among MSM. AIDS Educ Prev. 2004 Oct;16(5):448-58. doi: 10.1521/aeap.16.5.448.48739. PMID 15491956
- [Background] Marmor M, Penn A, Widmer K, Levin RI, Maslansky R. Coronary artery disease and opioid use. Am J Cardiol. 2004 May 15;93(10):1295-7. doi: 10.1016/j.amjcard.2004.01.072. PMID 15135709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: Sept. 2002 - March 2004. High-risk, HIV-seronegative, New York City men who have sex with men (MSM) were informed of the study by field workers at MSM-oriented bars, clubs and community events; advertisements in magazines distributed at such venues; and e-mails to persons offering sexual services for MSM on the Internet.
Groups:
- Placebo: Participants in this arm received placebo.
Period: Enrollment (Month 0)
Arm/Group | Bupropion | Placebo
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0
Period: Month 3
Arm/Group | Bupropion | Placebo
Started | 20 | 21
Completed | 16 | 18
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Period: Month 6
Arm/Group | Bupropion | Placebo
Started | 16 | 18
Completed | 16 | 17
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Month 9
Arm/Group | Bupropion | Placebo
Started | 16 | 17
Completed | 15 | 14
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Median (Full Range); unit: years] | 32.5 [23 to 48] | 32 [20 to 48] | 32 [20 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 10 | 16 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: The Number of Sexual Partners in Unprotected Anal Intercourse Reported at 6 Months Minus the Number Reported at Enrollment.
Description: The self-reported number of partners in unprotected anal intercourse during the 3 months prior to interview as reported at the Month 6 visit minus reported at the enrollment visit.
Time Frame: Enrollment to Month 6
Population: Subjects remaining in study through 6-Month study visit.
Measure: Median (Full Range); unit: Sexual partners
Groups:
- Bupropion; Placebo: 6 months
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 16 | 17
Sexual partners | -2.5 [-50 to 0] | -4 [-10 to 4]
Statistical Analysis 1: Comparison: Bupropion vs Placebo; Test type: Superiority or Other; p = 0.9, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.5

2. Secondary Outcome: Change in the Frequency Per Month of Use of Recreational Drugs Between Enrollment and Month 6 Measured by Questionnaire.
Description: Within-individual changes in the frequency of use of recreational drugs per month in the 3 months prior to interview reported at the Month 6 visit minus that reported at the enrollment visit.
Time Frame: Month 6 compared to Month 0 (enrollment)
Population: All subjects who were randomized, met study inclusion/exclusion criteria and were followed through Month 6
Measure: Median (Full Range); unit: Drug-using occasions per month
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 16 | 17
Drug-using occasions per month | 0.5 [-7.5 to 23] | 0 [-15 to 15]
Statistical Analysis 1: Comparison: Bupropion vs Placebo; Wilcoxon rank test; Test type: Superiority or Other; p = 0.3, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.5

3. Secondary Outcome: Incidence of Sexually Transmitted Infections Between Study Entry and Month 6 (Measured by Questionnaire and Laboratory Testing)
Description: Number of participants with incident sexually transmitted disease between enrollment the Month 6 interview.
Time Frame: Enrollment to Month 6
Population: Self-reported and laboratory identified sexually transmitted infections
Measure: Number; unit: participants
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 21
participants | 3 | 1
Statistical Analysis 1: Comparison: Bupropion vs Placebo; Comparison of cumulative incidence proportions; Test type: Superiority or Other; p = 0.3, Fisher Exact; Risk Ratio (RR) = 3.15, 95% CI 2-sided [0.4 to 27.8]

4. Secondary Outcome: Change in Beck Depression Inventory - II (BDI-II) Scores Between Enrollment and Month 6.
Description: The BDI-II is a self-administered, multiple-choice questionnaire inquiring into the presence and severity of symptoms associated with depression. BDI-II scores range from 0 to 63, with 10-19 interpreted as mild-to-moderate; 20-29 as moderate-to-severe, and ≥ 30 as severe depression. The study outcome measure was the BDI-II score at Month 6 minus the BDI score at enrollment
Time Frame: Month 6 compared to enrollment (Month 0)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 16 | 17
units on a scale | -11.5 [-31 to 8] | -9 [-19 to 5]
Statistical Analysis 1: Comparison: Bupropion vs Placebo; Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.5

ADVERSE EVENTS:
Time Frame: From enrollment through the 9-month follow-up.
Arm/Group | Bupropion | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/21
Other Adverse Events (participants affected / at risk) | 18/20 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=20) | Placebo (N=21)
Hospitalization with acute HIV infection (Infections and infestations) | 1 (1) | 0 (0) — Note that both SAEs occurred in a single individual enrolled in the bupropion arm of the study.
Hospitalization with left-sided chest pain radiating the left arm (General disorders) | 1 (1) | 0 (0) — Note that both SAEs occurred in a single individual enrolled in the bupropion arm of the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Bupropion (N=20) | Placebo (N=21)
Elevated diastolic pressure (>= 80 mm Hg) at Months 3, 6 or 9 (Cardiac disorders) | 10/16 (16) | 6/14 (10)
Elevated systolic pressure (>= 140 mm Hg) at Months 3, 6 or 9 (Cardiac disorders) | 2/16 (2) | 3/17 (4)
Weight loss (General disorders) | 0 (0) | 2 (2)
Dry mouth (General disorders) | 5 (8) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 5 (8)
Insomnia (Nervous system disorders) | 7 (11) | 0 (0)
Headache (Nervous system disorders) | 6 (10) | 4 (6)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4)
Agitation (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Fatigue (Nervous system disorders) | 5 (5) | 2 (2)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (11)
Sinus problem (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (7) | 1 (1)
Excessive sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Fever (Infections and infestations) | 1 (1) | 2 (2)
Chlamydia trachomatis infection (Infections and infestations) | 2 (2) | 1 (1)
Streptococcal infection of throat (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (6) | 9 (13)
Eye infection (Infections and infestations) | 3 (3) | 2 (2)
Heart palpitations (Cardiac disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
We achieved substantially lower recruitment than needed to adequately test the study hypothesis. We also experienced substantial losses-to-follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less